CLINICAL TRIAL: NCT04259476
Title: Low Dose Perioperative Ketamine Infusion and it's Effect on Postoperative Pain Score, Sedation Score and Narcotic Consumption in Patients Undergoing Spine Surgery: A Prospective Randomized Double Blind Control Trial.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Services Institute of Medical Sciences, Pakistan (Other Government)
Responsible Party: Principal Investigator, dr. sana siddiq, assistant professor, Services Institute of Medical Sciences, Pakistan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: servicesanesthesia
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2020-02-06 (Actual); Status verified 2020-02

CONDITIONS: for Post-operative Pain Relief in Spine Surgeries
Keywords: post-operative analgesia, ketamine, multi-modal therapy
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: randomized control trial
Who Masked: Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Active Comparator): WIll be given low dose perioperative ketamine infusion, as well as a ketamine bolus at start of surgery.
  Interventions: Drug: Ketamine Hydrochloride
- group B (Placebo Comparator): will be given normal saline infusion and bolus at start of surgery.
  Interventions: Drug: Ketamine Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — low dose perioperative ketamine infusion. and its effects on post-operative pain.
  Other Names: placebo, normal saline intrathecally.

SUMMARY:
Low dose perioperative ketamine infusion and it's effect on postoperative pain score, sedation score and narcotic consumption in patients undergoing spine surgery: A prospective randomized double blind control trial.

DETAILED DESCRIPTION:
Low dose perioperative ketamine infusion and it's effect on postoperative pain score, sedation score and narcotic consumption in patients undergoing spine surgery: A prospective randomized double blind control trial.

INTRODUCTION:

Recent advances in pain management advoctes the use of multimodal approach for post-operative pain therapy, as it reduces the side effects of individual drugs and attenuate pain responses at various sites in painpathways.. 6 if pain is not sufficiently managed, it can lead to various post-surgical complications and chronic pain..4 opiods are one of the commonly used drugs for provision of balanced anaesthesia as well as analgesia in the post surgical period. The use of opioids lead to various side effects, acute tolerance and hefty financial constraints if used in larger doses. In Pakistan, easy availability of narcotics also cause difficulty in choice of analgesics in post-operative pain.3 Ketamine , a phencyclidine derivative and dissociative anesthetic agent can cause significant analgesia when used in subanesthetic doses..1 it possess centrally mediated analgesic potential without any significant effect on patient's wakefulness and perception in dose of ≤0.3 mg/kg IV.2 Consensus guidelines on the use of intravenous ketamine for acute pain management from the American Society of Regional Anaesthesia and Pain Medicine, the American Academy of Pain Medicine and the American Society of Anaesthesiologists 2018 supports the use of sub anesthetic bolus dose of ketamine up to 0.35 mg/kg and infusions up to 1 mg/kg/hour for acute pain as adjuncts to opioids for perioperative analgesia.1 Low-dose IV ketamine infusion decrease opioid requirement by 40%. It also decreases pain scores, but these findings are less clear. No significant adverse effects have been reported with low-dose IV infusion of ketamine when used up to 48 hours after surgery5 We conducted this study to evaluate the effects of perioperative sub-anesthetic ketamine infusion, when continued in the post-operative period for 24 hours, on post-operative pain and sedation scores, overall narcotic and analgesics comsumptions and side effects in patients undergoing spine surgery in local population. Literature review did not show any such study conducted in Pakistan till date, results of this study can help innovate strategies of multimodel analgesia In local population.

Onjective:

The main objective of this study is to compare the effects of perioperative low dose ketamine infusion on postoperative pain , sedation score, adverse effects and total analgesics consumption in a placebo-controlled design Hypothesis Perioperative low dose ketamine infusion decreases the visual analogue score and total analgesic consumption without profound side effects in the study group.

Materials and Methods:

Study design: single blind prospective randomized control trial. Setting: After approval from ethical committee, this study will be conducted at the Department Of Anesthesiology and Surgical Intensive Care Uni t , services Hospital Lahore.

Duration of study: The proposed study will be completed in six months after approval of synopsis from services institute of medical sciences.

Sample size calculation:

Sample size is calculated by taking mean numeric pain rating score at 24 hours7 For ketamine group value NPRS is : 2.7±0.5 For control group NPRS value is : 3.1±1.0 Taking 95% Confidence interval level, 80 percent power of study and 5% alpha error sample size is calculated to be 60, taking 30 patients in each group.

Methodology:

This study will be conducted at services hospital lahore after institutional review board approval. After taking approval from review board, written informed consent will be taken from all the participants.

A total of 60 adult patients aged between 18 and 60 years old with American Society of Anesthesiology (ASA) physical status I-II scheduled for elective spine surgery will be allocated into two groups of 30 patients each. Regarding provision to maintain privacy, all participants' names will be concealed and replaced by code numbers to maintain privacy. Inclusion criteria included patients with ASA class I or II. Exclusion criteria included the following: BMI more than 40 kg/m2; poorly controlled arterial hypertension (blood pressure higher than 140/90 mmHg); respiratory, liver or kidney disease; and heart disease (heart block or myocardial ischemia).

During preanesthesia assessment, patients will be explained about the visual analogue scale (VAS) of 0-10 with 0 being "no pain" and 10 being "worst possible pain".

Patients will be randomly divided into two groups of 30 each by a sealed envelope technique.

Group A will be administered a bolus of intravenous ketamine of 0.25 mg/kg followed by an infusion of ketamine at a rate of 0.15 mg/kg/h.

Group B will be given a normal saline bolus and infusion at the same volume and rate.

The administration of bolus dose followed by infusion of both ketamine or saline will be started before the skin incision. The infusion (Mindray SK-500, Germany) will be continued intraoperatively and will be stopped after the skin closure but before the extubation of the patient. In order to avoid bias the medical staff who will not be involved in anesthetizing the patients will prepare the study drugs. The drugs will be prepared in 20 mL syringe (concentration of ketamine was 10 mg/ml), the saline syringes will also be labelled like ketamine syringes. Preoperatively the patients will be kept nil per oral for 6 hours before the surgery. Continuous monitoring of pulse, oxygen saturation, electrocardiogram, noninvasive blood pressure and end tidal carbon dioxide will be done perioperatively (Operon OM-12, Germany). The anesthesiologist administering anesthesia will not be aware of the group to which the patients belonged. The blood pressure will be monitored every 3 minutes. An 18 G IV line will be secured for drug administration and IV fluid management. IV glycopyrrolate 200 µg and IV metaclopramide 10 mg will given to all the patients as a premedication. IV induction will be done with propofol 2mg/kg and nalbuphine 0.1mg/kg. IV atracurium 0.5mg/kg will be used for endotracheal intubation. Maintenance of anesthesia will continue with sevoflurane and 100% oxygen. Fluid management will be done with IV ringer lactate. The reversal of the residual neuromuscular blockade will be done with IV neostigmine 0.05 mg/kg and glycopyrrolate 0.02 mg/kg. Endotracheal tube will be removed on complete recovery of the airway reflexes. The individual involved in data collection of pain scores will not be aware of the group to which the patient belonged. Similarly, the staff who provided the postoperative care in the hospital were unaware of the patient group. The patients will transferred to the post anesthesia care unit (PACU) and pain scores and sedation score will be noted on arrival, 1hr,3hr,6hr,8hr,12hr and 24 hr postoperatively using VAS and ramsey sedation scores respectively. The patients will be kept in post anesthesia care unit for 3 h. Patients will be shifted to the ward and will be given IV ketorolac 30 mg 12 hourly. All the patients who complained of pain score of VAS 4 or above will be provided provided rescue analgesia of IV nalbuphine bolus 0.1 mg/kg and time will be noted. The total amount of nalbuphine given in 24 h will be noted for both the groups. Side effects of ketamine and nalbuphine such as hallucination, sedation, nausea, vomiting and respiratory depression will be recorded. For hallucination IV haloperidol 5mg, for nausea and vomiting IV metoclopramide 10 mg and for respiratory depression (respiratory rate less than 9/min) IV naloxone will be given.

Data Analysis: The results will be analyzed using SPSS version 25.0.0 software (IBM. Results will be presented as mean ± standard deviation or as number of patients. Statistical significance of comparison of gender between two groups will be analyzed with Chi-square test. Statistical significance of age, weight, duration of surgery, VAS and nalbuphine consumption between two groups will be tested with independent sample t-test.

ELIGIBILITY:
Inclusion Criteria:

- A total of 60 adult patients aged between 18 and 60 years old with American Society of Anesthesiology (ASA) physical status I-II scheduled for elective spine surgery

Exclusion Criteria:

* BMI more than 40 kg/m2
* poorly controlled arterial hypertension (blood pressure higher than 140/90 mmHg)
* respiratory, liver or kidney disease
* heart disease (heart block or myocardial ischemia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
post operative pain score | upto 24 hours
  visual analogue scoring will be done for 24 hours post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- Services Institute of Medical Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No